CLINICAL TRIAL: NCT01907061
Title: Acute Renal Failure Post Liver Transplantation: The Role of Cytokines and Oxidative Stress
Brief Title: Acute Renal Failure Post Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 007-157
Record Dates: First submitted 2012-11-16; First posted 2013-07-24 (Estimated); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Acute Renal Failure
Keywords: acute renal failure; post liver transplant
MeSH Terms: conditions — Acute Kidney Injury | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 600 mg N-acetylcysteine or placebo IV (Active Comparator): 600 mg N-acetylcysteine or placebo IV perfused over 15 minutes during the transplant procedure, prior to reperfusion,
  Interventions: Drug: N-acetylcysteine; Drug: Placebo
- 600 mg N-acetylcysteine or placebo NG (Active Comparator): 600 mg NAC or placebo administered via NG tube starting at 12 hrs + 30 min post O.R. infusion,
  Interventions: Drug: N-acetylcysteine; Drug: Placebo
- N-acetylcysteine or placebo q 12 hour (Active Comparator): 600 mg NAC or placebo administered via NG tube every 12 hrs + 30 min for 3 additional doses (at 24, 36 and 48 hrs post O.R. infusion). The total administration will be 3000 mg over a 48 hr period.
  Interventions: Drug: N-acetylcysteine; Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — drug will be administered via IV,NG
  Other Names: NAC
Drug: Placebo — placebo or NAC will be given
  Other Names: Placebo in place of NAC

SUMMARY:
Trial to test the effect of administering N-acetylcysteine on cytokines and markers of oxidant stress and the incidence of acute renal failure post liver tranplant

DETAILED DESCRIPTION:
1. To determine levels of pro-inflammatory cytokines and oxidative stress markers in liver transplant patients during post-transplant period
2. To correlate changes in pro-inflammatory cytokines and markers of oxidative stress to acute renal failure and acute rejection
3. To determine the impact of using N-acetylcysteine on cytokines and markers of oxidative stress and the incidence of acute renal failure post liver transplantation

ELIGIBILITY:
Inclusion Criteria:

* First liver transplant
* Normal renal function before transplantation [serum creatinine ≤ 1.5 mg / dl]
* No requirements for dialysis before transplantation
* Age greater than 18 years

Exclusion Criteria:

* Re-transplant
* Renal dysfunction i.e. serum creatinine > 1.5 mg/dl
* Need for dialysis before transplantation
* Presence of Hepatorenal or Hepatopulmonary syndrome*
* Combined liver and kidney transplant
* Peptic ulcer disease
* Pregnancy

Ages: 18 Years to 71 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
To determine levels of pro-inflammatory cytokines and oxidative stress markers in liver transplant patients during post-transplant period | 6 months
  Cytokines in patients receiving N-acetylcysteine versus those receiving placebo during liver transplantation will be compared.

SECONDARY OUTCOMES:
To correlate changes in pro-inflammatory cytokines and markers of oxidative stress to acute renal failure and acute rejection | 6 months
  F2-isoprostanes levels in the two groups will be compared to evaluate the role in acute renal failure and acute rejection in patients recieving a liver transplant
iTo determine the impact of using N-acetylcysteine on cytokines and markers of oxidative stress and the incidence of acute renal failure post liver transplantation | 6 months
  N-acetylcysteine or placebo will be given to patients recieving a liver tranplant cytokines and oxidative stress markers will be compared between the two groups to determine if N-acetylcysteine will impact acute renal failure post liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Yousri M. Barri, MD, Principal Investigator — Baylor Health Care System
Locations (1):
- Annette C. and Harold C. Simmons Tranplant Institute at Baylor Medical Center Dallas, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No